CLINICAL TRIAL: NCT03881865
Title: P25/30 Somatosensory Evoked Potentials Are Associated With Neurological Prognosis of Comatose Survivors After Out of Hospital Cardiac Arrest
Brief Title: P25/30 SSEPs and Neurological Prognosis After Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18/P/088
Record Dates: First submitted 2018-11-19; First posted 2019-03-20 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-04

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Somatosensory Evoked Potential; cardiac arrest; prognosis; P25/30
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Title:

Early recorded P25/30 somatosensory evoked potentials are associated with neurologic prognosis of comatose survivors after out of hospital cardiac arrest.

Design:

Prospective, observational, non-interventional, study - prospective collection of data and interpretation. Analysis of the data and assessment of prognostic value of the P25/30 in critically ill patients post cardiac arrest.

Study Aims:

To be the first attempt to validate the prognostic potential of early recording [between 24-36 hours post Return Of Spontaneous Circulation] of P25/30 potentials in comatose survivors who are admitted to a British Intensive care unit after out of hospital cardiac arrest and who are not treated by hypothermic targeted temperature management.

[Validation of the prognostication significance of P25/30 Somatosensory Evoked Potentials in predicting neurologic outcome in comatose survivors post out of hospital cardiac arrest].

Outcome Measures:

Primary Endpoint: Neurologic outcome assessed by Cerebral Performance Category score at hospital discharge.

Secondary endpoints: Mortality at hospital discharge and 28 days [which occurs first], comparison of prognostic benefit of N20 and P25/30 based multimodal prognostic models.

Population:

Comatose survivors, after out of hospital cardiac arrest, treated in Derriford Hospital ICU, Penrose and Pencarrow wards.

Eligibility:

Adults [>18 years old], out of hospital cardiac arrest, comatose after Return Of Spontaneous Circulation, admission to intensive care Estimated Duration:36 months

DETAILED DESCRIPTION:
Recruitment and Conduction: In the first 24 hours in the Intensive Care Unit [ICU] the patients will be assessed for eligibility. If they meet the inclusion criteria, their Next Of Kin will be approached by a member of the study team. An explanation of the study design, the study protocol and the study objectives, as well as a specific relative information sheet for the study, will be provided. Meeting with the NOK is done ideally before the SSEP [SomatoSensory Evoked Potentials] recording or, in case of non-availability of the Next of kin, after the SSEP recording. The next of kin will have at least 24 hours to decide whether or not to participate in the study.

N20 and P25/30 SSEP are expected to be recorded and then during the study interpretation of the results the presence or absence of either or both with the neurological outcome will be assessed The SSEP recording as a prognostication adjunct after out of hospital cardiac arrest is part of the usual, established Derriford ICU policy for the management of the comatose survivors after out of hospital cardiac arrest and is not added or at any way modified, because of the study. The study purpose is the interpretation of the recording sheet of the SSEP test in order to answer the question whether the P25/30 potential that is recorded along with the N20 may have prognostic significance for the patients' neurological outcome. SSEPs must be recorded between 24-36 hours after ROSC [Return of Spontaneous Circulation]. Mild to moderate hypothermia ≥35 does not abolish the cortical N20 responses. Median or ulnar nerve bilaterally will be stimulated. Cortical N20 and P25/30 response is to be described as bilaterally absent (which is a good predictor of poor neurological outcome), or in other cases in may be present on one or both sides. If the cortical N20 response is absent, the presence of the peripheral N9 and N13 response must be present to ensure that the response has arrived at the cortex. Cervical lesions need to be excluded if Cortical N20 response is absent. After the SSEP recording, for those patients who informed consent is obtained from their next of kins and are enrolled to the study, a copy of each recording will be produced for the study purposes by one member of the study team who is not participating in the interpretation of the recording. This copy will be anonymised by giving a specific number for the study. After that, the anonymised copy will become available to the first and to the second interpreter [both members of the study team (neurophysiology)] who will interpret the recordings with regards to the presence and absence of the N20 and P25/30 SSEPs and they will record the results of their interpretation in the results databank. The two interpreters will be blinded for the personal and the clinical details of the patient. Also each one of the interpreters will not be aware about the result of the interpretation of the other. The ICU clinicians will not be aware about the results of the P25/30 interpretation as this will be part of the study and should not be disclosed to them during the conduction of the study. In this way, the P25/30 interpretation results will be impossible to affect the treatment of the patients and / or any of the clinical decisions made about them by the ICU clinicians. In the unlikely event that there was a discrepancy in interpretation of the SSEP recording between the two delegated interpreters, then a third member [not a member of the study team] of the Neurophysiology team would be asked to review the anonymised recording only in order to decide about the result. As the P25/30 pottential could be generated in the absence of N20 as they come from two distinct areas of the brain cortex, the presence of either the P25/30 or the N20 would be confirmed when the amplitude of each one is equal or higher than the amplitude threshold [0.5 microvolts] used for the analysis of the SSEPs. The presence and the amplitude of P25/30 will not be dependent on the presence of N20 in the same recording as each one of them can exist in the absence of the other. Measurement of the amplitude of recorded P25/30 and N20 and their combinations. Test if there is a correlation of the recorded amplitudes and their ratio [P25/30 to N20] with the positive predictive value of N20 for the favourable neurological outcome. After the SSEP recording has been conducted, between 24 and 36 hours post ROSC, the patients will be followed up by members of the study team. Those members of the team will assess the patients, by Cerebral Performance Category and full neurologic clinical examination, on the day of ICU discharge and on the day of their discharge from Derriford Hospital. The online system SALUS of Derriford hospital will be used to follow up the patients after their discharge from ICU and before their discharge from the hospital. The neurologic outcome, assessed with the Cerebral Performance Category [CPC], will be recorded. If a study participant died on ICU as a result of severe brain dysfunction or after the decision of ICU Consultant to be withdrawn from invasive organ support due to extremely poor prognosis, the discharge CPC would be the most recently recorded, after the patient have remained consistently off sedation [for a period of time varied for different sedatives or combination of sedatives]. If a participant died unexpectedly from another cause rather than severe brain dysfunction, then the most recent CPC before death [if available] will be recorded as indicative of neurologic outcome for the patients. In case the CPC could not be assessed, the patient would be excluded from the study analysis. The Results of the CPC assessment and the outcome of the patients will be stored in the general study databank for further analysis. At the End of the study, all data will be merged and statistically analysed and from the result of this analysis one or more relevant manuscripts must be submitted to a peer-review journal within the first 4 months after the completion of the study. For each one of the patients-participants, the following clinical data must be collected prospectively, during the conduction of the study [at different stages i.e. at the time of enrolment and follow up] and must be kept safely in an anonymised form in a suitable database. The principles of patients' confidentiality and privacy must be applied at all times. Age, Gender, Comorbidities, Pre-admission performance status [Assessed by the ECOG/WHO (Eastern Cooperative Oncology Group/World Health Organisation) performance status score, Cardiac Arrest Rhythm [Rhythm that was initially recorded after cardiac arrest, usually at scene], Bystander - witness of cardiac arrest and Cardiopulmonary resuscitation, Anoxic time [total time between cardiac arrest was noted and ROSC]. If multiple episodes of cardiac arrest then the sum of all anoxic times to be considered. GCS before intubation [total or with components if available]. Aetiology of cardiac arrest [cardiac or non-cardiac or unknown].CT [Computed Tomography] scan report if performed because it was clinically indicated.Cerebral performance category at ICU discharge and Hospital discharge. Date of death, number of days post ROSC that death occurred.ICU length of stay, hospital length of stay.Time of SSEP performed [hours post ROSC].Time between ROSC and ICU admission, First 24 hours post ROSC: mean SaO2 [arterial oxygen saturation], mean PaO2 [arterial partial pressure of oxygen], mean PaCO2 [arterial partial pressure of carbon dioxide], mean heart rate, mean blood pressure, mean Glucose levels, mean Lactate levels, mean pH, mean BE, Urea and Creatinine levels, liver function tests, Plasma sodium levels, Temperature, Sequential Organ Failure Assessment Score. No particulars tests needed for the study purposes.

The primary outcome measure is the CPC score at hospital discharge with discrete values ranging from 1 to 5. The score will be dichotomised as 1-2 (positive or good outcome) and 3-5 (negative or poor outcome). Sensitivity, specificity and predictive values of P25/30 in predicting poor outcome will be computed and the results compared to that of N20. Where appropriate, parameter estimates will be presented with 95% confidence intervals. Significant demographic and clinical predictors of poor neurological outcomes will be assessed and identified using regression models. Statistical data analysis will be undertaken once data collection from the required number of participants is completed. No interim analysis is scheduled for this study. Analyses will be performed in SPSS [Statistical Package for the Social Sciences] version 24 (or later). Sample size calculation was based on diagnostic test accuracy (adequate sensitivity) of P25/30. Previous studies on patients treated by hypothermic targeted temperature management showed that the sensitivity of P25/30 in predicting poor outcome is 90.12% (95% Confidence Interval, 81.5-95.6%). Though the proposed study will be based on those who are not treated by hypothermic targeted temperature management, the result (90%) is the 'best' available information regarding pre-determined sensitivity of P25/30. From experience of the team and analysis of the past three-years pilot data, the prevalence of poor outcome was assumed to be 75%. In order the maximum marginal error of estimate does not exceed from 5% with 95% confidence level, and adjusting for drop-out/lack of consent at 3%, the total required sample size will be 191. No power was assumed in the calculation of the sample size as there is no testing of hypothesis. Whenever applicable, a 5% level of significance will be used. As this is not an interventional study, the chance to terminate the trial is minimal. Spurious and/or missing data will be summarised and reasons for missingness given where possible. All data analyses will be based on the complete data only. Statistical analysis of the data will be performed at the end of the study. If deemed necessary, a separate statistical analysis plan (SAP) can be prepared prior to the completion of the study and approved by the oversight committee. The study team will discuss any deviation from the analysis plan and report it to the oversight committee. Any revisions to the SAP will be documented, including a brief justification and timing of revision. All eligible participants will be included in the analyses.

All the patients enrolled in the study are expected to be in coma at the time of enrollment. This is a reality about most of the ICU patients. Therefore, within the first 24 hours after ICU admission, the members of the study group will discuss with the next of kin of the patients regarding the potential participation in the study and the informed consent process. f the participants in the study regain full mental capacity to provide informed consent and make informed decisions after their enrollment in the study, then the participants will be fully informed about the study by a member of the study group and they will be asked if they agree to continue with their participation in the study. If the participants are happy to remain in the study cohort then their data will be used for analysis and publication purposes. If the participants decide anytime to withdraw from the study then their decision will be respected but it will be explained that that their data already collected may still be analysed as part of the study. The same options will be available for the next of kin that would have consented initially for the participation of patients in the study.

ELIGIBILITY:
Inclusion Criteria:

1. All adult comatose survivors after out of hospital cardiac arrest who are admitted to Derriford Hospital Intensive Care Unit [Penrose and Pencarrow wards]. The cause of cardiac arrest may be cardiac and/or non-cardiac or unknown at the time of enrolment.
2. All patients must be comatose before intubation [GCS equal or lower than 8].
3. All patients must be on one or more invasive organ support [e.g. Endotracheal intubation and mechanical ventilation, vasopressor and/or inotropic support, Continuous Renal Replacement Therapy Sedated and/or on neuromuscular blocking agents].
4. All patients must be sedated before and during the time of SSEP recording. If clinically indicated, neuromuscular blocking agents may also be used.
5. All patients must be on targeted temperature management as per Derriford ICU policy and protocol: For the first 24 hours after ICU admission, the target-temperature is 36°C with temperature control commencing within the first hour after critical care admission. For the next 48 hours the temperature of the patients will be maintained between 36-37°C. The aforementioned temperature targets are achieved with external cooling devices.
6. Patients must have a CT scan of the head if severe cerebral pathology which is part of the exclusion criteria is clinically suspected.
7. Absence of all exclusion criteria

Exclusion Criteria:

1. Non-comatose patients after ROSC
2. Coma secondary to Intracranial and Intracerebral haemorrhage
3. Patients with haemorrhagic shock
4. Patients with severe neurologic disability [CPC level higher than 2] during the pre-cardiac arrest period
5. Presence of active Demyelinating disease or past medical history of Demyelinating disease
6. Trauma-related Cardiac arrest
7. Previously or during the current admission diagnosed Spinal Cord and /or brain stem lesions
8. Patients with Implantable defibrillator device [incompatibility with SSEP recordings device]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult [> 18 years old] comatose survivors after non-trauma-related out of hospital cardiac arrest who are admitted to Derriford Hospital Intensive Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Cerebral Performance Category [CPC] score | up to 30 days after cardiac arrest
  Neurological status of the participants assessed by the use of CPC score. CPC has 5 different scores describing the neurological outcome. CPC score 1: Full recovery or mild disability CPC score 2: Moderate Disability but independent in activities of daily living CPC score 3: Severe disability - Dependent in activities of daily living CPC score 4: persistent vegetative state CPC score 5: Death CPC scores 1 and 2 are considered positive [good] neurological outcomes, whereas scores 3-5 are considered negative [poor] neurological outcomes.

SECONDARY OUTCOMES:
Mortality | up to 30 days after cardiac arrest
  Number of patients that died during the study period
Correlation between P25/30 somatosensory evoked potentials presence and favourable prognosis | Up to 30 days after cardiac arrest
  Number of patients in whom P25/30 were present and they had favourable neurologic outcomes [CPC scores 1 and 2]

CONTACTS AND LOCATIONS:
Overall Officials: Nikitas Nikitas, MD, PhD, Principal Investigator — University Hospitals Plymouth Department for Research Development and Innovation
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD to be shared via ClinicalTrials.gov
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Attached to ClinicalTrials.gov record
Access Criteria: ClinicalTrials.gov

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT03881865/Prot_SAP_001.pdf